CLINICAL TRIAL: NCT03645031
Title: Acute Intermittent Hypoxia and Breathing in Neuromuscular Disease
Acronym: AIH-ALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201801131; OCR18018 (Other: OnCore)
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS); Neuromuscular Diseases
Keywords: acute intermittent hypoxia (AIH); respiratory motor function; hypoxia; normoxia; EMG (electromyography)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neuromuscular Diseases; Hypoxia | interventions — Insemination, Artificial, Homologous

STUDY DESIGN:
Intervention Model Description: Participants will complete both the AIH and the sham AIH visits. The order of these visits will be randomized, but all subjects will complete both visits in the course of the study.
Who Masked: Participant
Masking Description: Participants will be blind to the order of the AIH/sham AIH visits, but this information will be provided to the participant after completion of last visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALS Group (Experimental): Participants will complete a single 45 minute session of acute intermittent hypoxia (AIH), as well as, the 45 minute sham AIH session, consisting of breathing air with normal oxygen levels. Breathing, muscle activity and heart activity will be monitored before, during and after both procedures.
  Interventions: Other: Acute Intermittent Hypoxia; Other: Sham Acute Intermittent Hypoxia
- Healthy Control Group (Experimental): Participants will complete a single 45 minute session of acute intermittent hypoxia (AIH), as well as, the 45 minute sham AIH session, consisting of breathing air with normal oxygen levels. Breathing, muscle activity and heart activity will be monitored before, during and after both procedures.
  Interventions: Other: Acute Intermittent Hypoxia; Other: Sham Acute Intermittent Hypoxia

INTERVENTIONS:
Other: Acute Intermittent Hypoxia — AIH entails continuous breathing as the level of oxygen in the air is decreased, then returned to normal. Participants will alternate between breathing normal air and breathing hypoxic air (air that has less oxygen). Participants will complete a single 45 minute session of acute intermittent hypoxia (AIH). Breathing, muscle activity and heart activity will be monitored before, during and after the procedure. The intervals will last 1 minute each.
  Other Names: AIH
Other: Sham Acute Intermittent Hypoxia — Participants will complete the sham acute intermittent hypoxia, consisting of a single 45 minute session of breathing air with normal oxygen levels. All aspects of this procedure will otherwise be the same as for the AIH procedure. Breathing, muscle activity and heart activity will be monitored before, during and after the procedure.
  Other Names: Sham AIH

SUMMARY:
This project seeks to investigate the effects of a single acute intermittent hypoxia (AIH) session on respiratory and non-respiratory motor function and EMG (electromyography) activity on patients with ALS (amyotrophic lateral sclerosis) and healthy controls.

DETAILED DESCRIPTION:
Most ALS patients survive less than 5 years after diagnosis, and the main cause of death is respiratory failure. The investigators are interested in the therapeutic potential of acute intermittent hypoxia (AIH) for individuals with neuromuscular diseases, such as ALS. More than two decades of research indicates AIH elicits meaningful respiratory and non-respiratory motor recovery. Acute intermittent hypoxia (AIH) consists of alternating periods of breathing mildly hypoxic (lowered oxygen concentration) and normoxic (normal oxygen concentration) air.

The investigators propose to study mechanisms of respiratory plasticity associated with a single presentation of mild AIH. The fundamental hypothesis guiding this proposal is that even a single AIH trial improves respiratory (and non-respiratory) motor function in ALS patients procedure. Participants will then be asked to breathe air with reduced oxygen for short periods of time, for a duration of 45 minutes. The activity of your muscles and your heart function will be monitored throughout the procedure.

ELIGIBILITY:
Inclusion Criteria:

* a healthy adult
* clinical diagnosis of ALS
* baseline FVC >60% predicted for age, sex and height.

Exclusion Criteria:

* pregnant
* diagnosed cardiovascular disease
* a BMI >35 kg/m2
* currently take selective serotonin reuptake inhibitors (SSRI)
* history of seizures
* history of hospitalization for sepsis
* respiratory infection or took antibiotic medications within the past 4 weeks
* use external respiratory support during any waking hours
* participate in a pharmaceutical trial to treat ALS
* have any other medical condition the PI or medical director identify would make it unsuitable to participate.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara K Smith, PT, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UF Clinical Research Center, Gainesville, Florida
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ALS Group - AIH Followed by Sham; Healthy Control Group - AIH Followed by Sham Hypoxia: Participants will complete a single 45 minute session of acute intermittent hypoxia (AIH) as well as, the 45 minute sham AIH session, consisting of breathing air with normal oxygen levels two weeks later. Breathing, muscle activity and heart activity will be monitored before, during and after both procedures.
  Acute Intermittent Hypoxia: AIH entails continuous breathing as the level of oxygen in the air is decreased, then returned to normal. Participants will alternate between breathing normal air and breathing hypoxic air (air that has less oxygen). Participants will complete a single 45 minute session of acute intermittent hypoxia (AIH). Breathing, muscle activity and heart activity will be monitored before, during and after the procedure. The intervals will last 1 minute each.
  Sham Acute Intermittent Hypoxia: Participants will complete the sham acute intermittent hypoxia, consisting of a single 45 minute session of breathing air with normal oxygen levels. All aspects of this procedure will otherwise be the same as for the AIH procedure. Breathing, muscle activity and heart activity will be monitored before, during and after the procedure.
- ALS Group, Sham Followed by AIH; Healthy Control Group, Sham Followed by AIH: Participants will complete a single 45 minute session of sham intermittent hypoxia consisting of breathing air with normal oxygen levels, as well as a single 45 minute session of acute intermittent hypoxia (AIH) two weeks later. Breathing, muscle activity and heart activity will be monitored before, during and after both procedures.
Period: Overall Study
Arm/Group | ALS Group - AIH Followed by Sham | Healthy Control Group - AIH Followed by Sham Hypoxia | ALS Group, Sham Followed by AIH | Healthy Control Group, Sham Followed by AIH
Started | 7 | 8 | 8 | 6
Completed | 6 | 6 | 8 | 4
Not Completed | 1 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Patients with an ALS diagnosis and age matched healthy controls.
Groups:
- Total: Total of all reporting groups
Arm/Group | ALS Group | Healthy Control Group | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 7 | 7 | 14
Age, Continuous [Mean (Full Range); unit: years] | 65.3 [56 to 72] | 67.4 [60 to 75] | 66.2 [56 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 10 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 8 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 10 | 23
Vital capacity (% predicted) [Mean (Full Range); unit: Percentage] | 83.3 [61 to 113] | 105.2 [86 to 132] | 92.8 [61 to 132]
Amyotrophic Lateral Sclerosis Functional Rating Scale- Revised (ALS-RFS-R) [Mean (Full Range); unit: units on a scale] — The ALS-FRS-R is a scale that reflects the functional impact of ALS. The score consists of 12 subsections each rated on scale from 0-4. The subsections include speech, salivation, swallowing, handwriting, feeding, dressing/hygiene, walking, climbing stairs, dyspnea, orthopnea, and respiratory insufficiency. The total score was reported and is the sum of the 12 subsections (0-48 points) where higher scores represent more preserved function. Population: The healthy controls do not have an ALS-FRS score.
  units on a scale
    number analyzed (Participants) | 13 | 0 | 13
    (all) | 38.8 [33 to 45] |  | 38.8 [33 to 45]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Maximal Inspiratory Pressure (MIP)
Description: MIP is a maximal voluntary static contraction of the inspiratory muscles against a closed valve, measured at the mouth. The test will be repeated until 3 measurements are obtained within 10% variability and an average of the three trials is reported. The change in MIP will be the percent difference in pressure between the averaged baseline MIP and the averaged follow-up measure, which is tested 60 minutes after the gas intervention.
Time Frame: 3 Hours
Population: Individuals with an ALS diagnosis and age matched healthy controls.
Measure: Mean (Standard Error); unit: percentage change in MIP from baseline
Arm/Group | ALS Group | Healthy Control Group
Number analyzed (Participants) | 13 | 10
percentage change in MIP from baseline
  Sham Hypoxia | 0.3 (2.9) | -3.1 (2.3)
  AIH | -4.8 (1.6) | -5.0 (3.2)

2. Primary Outcome: Percent Change in Maximal Voluntary Grip Force
Description: Maximal static voluntary handgrip contractions will be evaluated in a seated position with the arm at the side and elbow flexed to 90 degrees. The test will be repeated until 3 measurements are obtained within 10% variability and then averaged. The change in grip will be the percent difference in force between the averaged baseline grip and the averaged follow-up grip measure, which is tested 60 minutes after the gas intervention.
Time Frame: 3 Hours
Population: Individuals with an ALS diagnosis and age matched unaffected controls.
Measure: Mean (Standard Error); unit: percent change in grip forcfrom baseline
Groups:
- Unaffected Control Group: Participants will complete a single 45 minute session of acute intermittent hypoxia (AIH), as well as, the 45 minute sham AIH session, consisting of breathing air with normal oxygen levels. Breathing, muscle activity and heart activity will be monitored before, during and after both procedures.
  Acute Intermittent Hypoxia: AIH entails continuous breathing as the level of oxygen in the air is decreased, then returned to normal. Participants will alternate between breathing normal air and breathing hypoxic air (air that has less oxygen). Participants will complete a single 45 minute session of acute intermittent hypoxia (AIH). Breathing, muscle activity and heart activity will be monitored before, during and after the procedure. The intervals will last 1 minute each.
  Sham Acute Intermittent Hypoxia: Participants will complete the sham acute intermittent hypoxia, consisting of a single 45 minute session of breathing air with normal oxygen levels. All aspects of this procedure will otherwise be the same as for the AIH procedure. Breathing, muscle activity and heart activity will be monitored before, during and after the procedure.
Arm/Group | ALS Group | Unaffected Control Group
Number analyzed (Participants) | 13 | 10
percent change in grip forcfrom baseline
  AIH | -8.2 (0.26) | -11.2 (0.24)
  SHAM | 14.5 (0.11) | 18.2 (0.07)

3. Primary Outcome: Percent Change in Sniff Nasal Inspiratory Pressure
Description: Maximal voluntary contractions of the inspiratory muscles measured with a pressure sensor placed in the nare. The test will be repeated until 3 measurements are obtained within 10% variability and then averaged. The change in sniff nasal inspiratory pressure will be the percent difference in pressure between the averaged baseline sniff nasal inspiratory pressure and the averaged follow-up measure, which is tested 60 minutes after the gas intervention.
Time Frame: 3 Hours
Population: Individuals with an ALS diagnosis and age matched healthy controls.
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Arm/Group | ALS Group | Healthy Control Group
Number analyzed (Participants) | 13 | 10
Percent Change from Baseline
  Sham | 2.5 (4.1) | 7.4 (5.9)
  AIH | 4.9 (5.0) | 5.8 (5.5)

4. Secondary Outcome: Percent Change in Minute Ventilation
Description: Minute ventilation is measured using a pneumotachograph connected to the face mask to record breath-by-breath volume and breathing rate, which is then multiplied to calculate minute ventilation. After achieving a stable tidal volume, 5 minutes of resting minute ventilation will be recorded and then averaged. The change in minute ventilation will be the percent difference in volume between the averaged baseline ventilation and the averaged follow-up ventilation, which is tested 60 minutes after the gas intervention.
Time Frame: 3 Hours
Population: Individuals with an ALS diagnosis and age matched controls.
Measure: Mean (Standard Error); unit: percentage change from baseline
Arm/Group | ALS Group | Healthy Control Group
Number analyzed (Participants) | 13 | 10
percentage change from baseline
  Sham hypoxia | 5.7 (7.3) | -5.6 (5.4)
  AIH | 19.5 (6.0) | 2.6 (7.2)

5. Secondary Outcome: Occlusion Pressure (P0.1)
Description: P0.1 is measured with a pressure transducer connected to a face mask and represents the pressure generated against a transiently occluded airway in the first 0.1 sec of inspiration. The generated during this initial period of inspiration is resistant to learning or sensory bias and is considered a clinical estimate of inspiratory drive. Five measurements will be conducted and then averaged, with 5-15 un-occluded breaths between each P0.1 measurement. The averaged pressures at baseline and 60 minutes post-gas intervention will be reported and will be expressed in cm H2O.
Time Frame: 3 Hours
Population: Individuals with an ALS diagnosis and age matched healthy controls who completed a single exposure to acute intermittent hypoxia. P0.1 during sham hypoxia presentations were not collected due to an oversight by study staff and cannot be reported.
Measure: Mean (Standard Deviation); unit: cm H2O
Groups:
- ALS Group: In people diagnosed with ALS, P0.1 was evaluated in conjunction with a single 45 minute session of acute intermittent hypoxia (AIH), which entails continuous breathing as the level of oxygen in the air is decreased, then returned to normal. Participants alternate between breathing normal air and breathing hypoxic air (air that has less oxygen). Participants completed a single 45 minute session of acute intermittent hypoxia (AIH).
- Healthy Control Group: In unaffected control participants, P0.1 was evaluated in conjunction with a single 45 minute session of acute intermittent hypoxia (AIH), which entails continuous breathing as the level of oxygen in the air is decreased, then returned to normal. Participants alternate between breathing normal air and breathing hypoxic air (air that has less oxygen). Participants completed a single 45 minute session of acute intermittent hypoxia (AIH).
- ALS Group - Sham Hypoxia: People diagnosed with ALS, underwent a single 45 minute session of acute intermittent hypoxia (AIH), which entails alternating between breathing normal air and breathing sham hypoxia, which is also normal air. Participants completed a single 45 minute session of sham hypoxia.
- Control Group: Unaffected control participants underwent a single 45 minute session of acute intermittent hypoxia (AIH), which entails alternating between breathing normal air and breathing sham hypoxia, which is also normal air. Participants completed a single 45 minute session of sham hypoxia.
Arm/Group | ALS Group | Healthy Control Group | ALS Group - Sham Hypoxia | Control Group
Number analyzed (Participants) | 9 | 6 | 0 | 0
cm H2O
  Baseline | -0.80 (0.58) | -0.60 (0.41) |  |
  60 minutes post-AIH | -0.83 (0.72) | -0.47 (0.53) |  |

6. Secondary Outcome: Percentage Change in Respiratory EMG Vector Magnitude
Description: EMG vector magnitude represents the composite surface EMG activity expressed from eight respiratory muscles (bilateral scalene, sternocleidomastoid, 2nd parasternal, and 8th external intercostal/diaphragm). The vector magnitude was calculated for each participant from the root mean square (RMS) values from each EMG channel, as the square root of the sum of the individual squared EMG channel amplitudes.
Time Frame: 3 Hours
Population: Individuals with an ALS diagnosis and age matched controls.
Measure: Mean (Standard Error); unit: percentage change from baseline
Arm/Group | ALS Group | Healthy Control Group
Number analyzed (Participants) | 13 | 10
percentage change from baseline
  Sham hypoxia | -24.5 (4.1) | 7.4 (13.1)
  AIH | 179.8 (45.9) | 352.3 (99.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from subject consent through 1 week following the last study visit. This timeframe is approximately 6 weeks.
Description: Adverse event definitions were consistent with clinicaltrials.gov definitions. Participants were asked at the beginning and end of every study visit to report any signs, symptoms, or occurrence that has occurred since their last encounter. Additionally, a final assessment was conducted by phone, approximately one week after the last study visit.
Groups:
- ALS- AIH Group: Participants will complete a single 45 minute session of acute intermittent hypoxia (AIH), as well as, the 45 minute sham AIH session, consisting of breathing air with normal oxygen levels. Breathing, muscle activity and heart activity will be monitored before, during and after both procedures.
  Acute Intermittent Hypoxia: AIH entails continuous breathing as the level of oxygen in the air is decreased, then returned to normal. Participants will alternate between breathing normal air and breathing hypoxic air (air that has less oxygen). Participants will complete a single 45 minute session of acute intermittent hypoxia (AIH). Breathing, muscle activity and heart activity will be monitored before, during and after the procedure. The intervals will last 1 minute each.
- Healthy Control- AIH Group: Participants will complete a single 45 minute session of acute intermittent hypoxia (AIH), as well as, the 45 minute sham AIH session, consisting of breathing air with normal oxygen levels. Breathing, muscle activity and heart activity will be monitored before, during and after both procedures.
  Acute Intermittent Hypoxia: AIH entails continuous breathing as the level of oxygen in the air is decreased, then returned to normal. Participants will alternate between breathing normal air and breathing hypoxic air (air that has less oxygen). Participants will complete a single 45 minute session of acute intermittent hypoxia (AIH). Breathing, muscle activity and heart activity will be monitored before, during and after the procedure. The intervals will last 1 minute each.
  Sham Acute Intermittent Hypoxia: Participants will complete the sham acute intermittent hypoxia, consisting of a single 45 minute session of breathing air with normal oxygen levels. All aspects of this procedure will otherwise be the same as for the AIH procedure. Breathing, muscle activity and heart activity will be monitored before, during and after the procedure.
- ALS- SHAM GROUP; Healthy Control- SHAM Group: Participants will complete a single 45 minute session of acute intermittent hypoxia (AIH), as well as, the 45 minute sham AIH session, consisting of breathing air with normal oxygen levels. Breathing, muscle activity and heart activity will be monitored before, during and after both procedures.
  Sham Acute Intermittent Hypoxia: Participants will complete the sham acute intermittent hypoxia, consisting of a single 45 minute session of breathing air with normal oxygen levels. All aspects of this procedure will otherwise be the same as for the AIH procedure. Breathing, muscle activity and heart activity will be monitored before, during and after the procedure.
Arm/Group | ALS- AIH Group | Healthy Control- AIH Group | ALS- SHAM GROUP | Healthy Control- SHAM Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/11 | 0/14 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/11 | 0/14 | 0/11
Other Adverse Events (participants affected / at risk) | 2/14 | 1/11 | 4/14 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALS- AIH Group (N=14) | Healthy Control- AIH Group (N=11) | ALS- SHAM GROUP (N=14) | Healthy Control- SHAM Group (N=11)
Cough and sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Wrist sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shingles (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT03645031/Prot_SAP_000.pdf